CLINICAL TRIAL: NCT00174369
Title: Phase 2 Study Of The MEK Inhibitor PD-0325901 In Patients With Advanced Non-Small Cell Lung Cancer
Brief Title: MEK Inhibitor PD-325901 To Treat Advanced Non-Small Cell Lung Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Terminated [See Detailed Description for Termination Reason.]
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A4581002
Record Dates: First submitted 2005-09-09; First posted 2005-09-15 (Estimated); Last update posted 2009-03-17 (Estimated); Status verified 2009-02

CONDITIONS: Carcinoma, Non-Small-Cell Lung
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — mirdametinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- PD0325901 (Experimental): 15 mg BID
  Interventions: Drug: PD-0325901

INTERVENTIONS:
Drug: PD-0325901 — 15 mg BID

SUMMARY:
MEK is a critical member of the MAPK pathway involved in growth and survival of cancer cells. PD-325901 is a new drug designed to block this pathway and kill cancer cells. The purpose of this study is to study the effectiveness of PD-325901 in patients with non-small cell lung cancer. PD-325901 will be given by mouth as a pill twice a day, CT scans will be done and biopsies of a tumor and a blood sample will be taken before treatment to examine the how genes affect tumor response to the study medication. Blood samples will be taken to measure the amount of drug in the blood.

DETAILED DESCRIPTION:
This study was terminated prematurely on 23 March 2007 due to safety issues (ocular and neurological toxicity observed in another PD-0325901 study, A4581001) as well as lack of objective responses

ELIGIBILITY:
Inclusion Criteria:

* Histologically documented non-small cell lung cancer with metastases (Stage IV or recurrent disease) or locally advanced (Stage IIIB) with malignant pleural effusion with no expectation of further effects of prior anticancer therapy, and resolution of all acute toxic effects
* Adequate renal, liver, and bone marrow function, determined within 2 weeks prior to the first treatment and an ECOG status of <=1.
* Must have evidence of progression of disease within 6 months of most recent prior systemic anticancer therapy.

Exclusion Criteria:

* No parathyroid disorder or history of malignancy associated hypercalcemia
* No ongoing radiation therapy or radio-cytotoxic therapy within prior 4 weeks; No immunotherapy, biologic therapy, hormonal, or molecular targeted therapy within prior 2 weeks
* No concurrent serious infection or life-threatening illness (unrelated to tumor)
* No history of a malignancy (other tha non-small cell lung cancer) except those treated with curative intent for skin cancer (other than melanoma) or in situ breast or cervical cancer or those treated with curative intent for any other cancer with no evidence of disease for 5 years.
* No active seizure disorders or untreated brain metastases.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2005-11; Primary Completion 2007-06 (Actual); Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
To determine the activity of PD-0325901 in advanced non-small cell lung cancer | Duration of trial

SECONDARY OUTCOMES:
To determine the progression-free survival | Duration of trial
To determine the duration of response | Duration of trial
To determine the overall survival | Duration of trial
To determine the safety profile of PD-0325901 | Duration of trial
To explore pharmacogenomic and cancer biomarkers (gene and/or protein expression profiling) relationships with cancer- and treatment-related outcomes duration of response | Duration of trial
To evaluate PD-0325901 population pharmacokinetics and explore its correlation with efficacy and safety parameters | Duration of trial
To explore pharmacogenomic and cancer biomarkers (gene and/or protein expression profiling) relationships with cancer- and treatment-related outcomes | Duration of trial

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (13):
- United States (13):
  - Pfizer Investigational Site, Greenbrae, California
  - Pfizer Investigational Site, La Jolla, California
  - Pfizer Investigational Site, San Diego, California
  - Pfizer Investigational Site, San Mateo, California
  - Pfizer Investigational Site, Tampa, Florida
  - Pfizer Investigational Site, Ann Arbor, Michigan
  - Pfizer Investigational Site, Detroit, Michigan
  - Pfizer Investigational Site, Farmington Hills, Michigan
  - Pfizer Investigational Site, Coon Rapids, Minnesota
  - Pfizer Investigational Site, Fridley, Minnesota
  - Pfizer Investigational Site, Robbinsdale, Minnesota
  - Pfizer Investigational Site, New York, New York
  - Pfizer Investigational Site, Philadelphia, Pennsylvania

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A4581002&StudyName=MEK%20Inhibitor%20PD-325901%20to%20Treat%20Advanced%20Non-Small%20Cell%20Lung%20Cancer